CLINICAL TRIAL: NCT00042497
Title: A Phase II, Multicenter, Open-Labeled Study of Immunotherapy With Autologous Dexosomes for Patients With Stage IV Melanoma
Brief Title: Immunotherapy With Autologous Dexosomes for Patients With Stage IV Melanoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Anosys (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AN2002-04
Record Dates: First submitted 2002-07-30; First posted 2002-08-01 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

INTERVENTIONS:
Biological: autologous dexosomes loaded with tumor-specific peptides

SUMMARY:
The objective is to determine the safety and efficacy of dexosome immunotherapy in patients with Stage IV malignant melanoma

ELIGIBILITY:
* Patients with Stage IV metastatic melanoma with 0-1 prior treatments for metastatic disease.
* All patients must have distant skin, subcutaneous, or nodal metastases (M1a) or lung metastases (M1b), measurable disease, normal lactate dehydrogenase levels, and HLA type A1, A2, or B35.
* Patients must have adequate organ function and an estimated life expectancy of at least 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-07